CLINICAL TRIAL: NCT02933970
Title: Stepped-Wedge Randomized Control Trial to Compare Integrated, Co-located, Telemedicine-based HCV Management for Individuals on Opiate Agonist Treatment Versus Usual Care Treatment of HCV of Individuals on Opiate Agonist Treatment
Brief Title: Comparison of Telemedicine to Usual Care for HCV Management for Methadone-maintained Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Talal (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Andrew Talal, Professor, State University of New York at Buffalo
Organization: State University of New York at Buffalo (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Telemedicine vs. Usual Care
Record Dates: First submitted 2016-09-24; First posted 2016-10-14 (Estimated); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Referral-HCV seropositive subjects enrolled for at least 12 months in an opiate agonist treatment (OAT) program will be referred to an off-site liver specialist
- Intervention (Other): Telemedicine - HCV seropositive subjects enrolled for at least 12 months in an OAT program will be treated on site by a liver specialist via two-way video conferencing. (telemedicine)
  Interventions: Other: Telemedicine

INTERVENTIONS:
Other: Telemedicine — Patients will be linked with the provider via two-way video-teleconferencing facilitated by an onsite OAT program staff member
  Other Names: Two way video conferencing
  Arms: Intervention

SUMMARY:
To compare the effectiveness of a patient-centered, opiate agonist treatment (OAT)-integrated telemedicine-based approach for management and delivery of hepatitis C virus (HCV) treatment to persons with substance use disorders (PWSUD) versus usual care, which we anticipate in most cases will be referral to an offsite location for HCV management. The effectiveness will be expressed through the primary patient centered and clinical outcome, achievement of viral eradication, defined as undetectable HCV RNA 12 weeks post-treatment cessation.

DETAILED DESCRIPTION:
The study is a non-blinded stepped wedge cluster randomized controlled trial with two arms: onsite HCV management through telemedicine versus HCV management through usual care, referral to an offsite hepatitis specialist (Referral). The arm assignment is at the cluster (clinic) level. After an initial period (9 months) in which all clinics implement the control intervention (usual care), at regular intervals (i.e., the "steps") of 9 months duration each, one group of clinics is randomized to cross over from the Usual Care arm to the Telemedicine arm. The process continues until all clinics have crossed over to implement telemedicine, and thus all clinics contribute data to both interventions. In addition, patients cured of HCV are followed for two years post-treatment cessation to assess for reinfection or relapse of HCV RNA.

ELIGIBILITY:
Inclusion Criteria:

1. HCV antibody detected
2. Ability and willingness of subject or legal representative to provide written informed consent.
3. 18 years of age
4. A minimum of 12-month enrollment in the opiate agonist treatment program
5. Likely to be adherent to the therapeutic regimen
6. Covered by medical insurance

Exclusion Criteria:

1. Mental instability or incompetence, such that the validity of the informed consent or ability to be compliant with the study is uncertain.
2. <18 years of age
3. < 12 months enrolled in an opiate agonist treatment program.
4. Non-compliance with therapeutic regimen defined as three consecutive missed appointments that will result in a discussion between the principal investigator at the site and the study participant to determine the reason for the missed appointments. Continuation in the study for the participant will be assessed on a case-by-case basis between the study PI and the site PI.
5. Lack of medical insurance coverage
6. Ineligibility for HCV treatment
7. Active treatment for HCV at the time of the study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Talal, MD, Principal Investigator — SUNY Buffalo
Locations (1):
- Andrew H Talal, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
At the completion of the study, the data will be filed with the Patient-Centered Outcomes Research Institute and will be publicly availability.

REFERENCES:
- [Derived] Talal AH, Markatou M, Zeremski M, Liu A, Dharia A, George SG, Taylor M, Davis K, Silber A, Brown LS, Tobin JN. Opioid treatment program-integrated facilitated telemedicine for hepatitis C treatment: a hybrid effectiveness-implementation analysis. BMC Complement Med Ther. 2025 Oct 15;25(1):377. doi: 10.1186/s12906-025-05138-9. PMID 41094463
- [Derived] Dickerson SS, George SJ, Ventuneac A, Dharia A, Talal AH. Care Integration for Hepatitis C Virus Treatment Through Facilitated Telemedicine Within Opioid Treatment Programs: Qualitative Study. J Med Internet Res. 2024 Jun 12;26:e53049. doi: 10.2196/53049. PMID 38865703
- [Derived] Talal AH, Markatou M, Liu A, Perumalswami PV, Dinani AM, Tobin JN, Brown LS. Integrated Hepatitis C-Opioid Use Disorder Care Through Facilitated Telemedicine: A Randomized Trial. JAMA. 2024 Apr 23;331(16):1369-1378. doi: 10.1001/jama.2024.2452. PMID 38568601
- [Derived] Ventuneac A, Dickerson SS, Dharia A, George SJ, Talal AH. Scaling and Sustaining Facilitated Telemedicine to Expand Treatment Access Among Underserved Populations: A Qualitative Study. Telemed J E Health. 2023 Dec;29(12):1862-1869. doi: 10.1089/tmj.2022.0534. Epub 2023 May 26. PMID 37252770
- [Derived] Talal AH, Sofikitou EM, Wang K, Dickerson S, Jaanimagi U, Markatou M. High Satisfaction with Patient-Centered Telemedicine for Hepatitis C Virus Delivered to Substance Users: A Mixed-Methods Study. Telemed J E Health. 2023 Mar;29(3):395-407. doi: 10.1089/tmj.2022.0189. Epub 2022 Aug 4. PMID 35925809
- See also: Related Info — http://www.who.int/mediacentre/factsheets/fs164/en/.
- See also: Related Info — http://www.cdnetwork.org/teamc

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Opioid Treatment Programs
Groups:
- Sequence 1: 27 Month Usual Care, 9 Months Telemedicine: 27 months of usual care: referral-HCV seropositive subjects enrolled for at least 6 months in an opiate agonist treatment (OAT) program will be referred to an off-site liver specialist.
  Then, 9 months of telemedicine: patients will be linked with the provider via two-way videoconferencing facilitated by an onsite case manager.
- Sequence 2: 18 Month Usual Care, 18 Months Telemedicine: 18 months of usual care: referral-HCV seropositive subjects enrolled for at least 6 months in an opiate agonist treatment (OAT) program will be referred to an off-site liver specialist.
  Then, 18 months of telemedicine: patients will be linked with the provider via two-way videoconferencing facilitated by an onsite case manager.
- Sequence 3: 9 Months of Usual Care Followed by 27 Months Telemedicine: 9 months of usual care: referral-HCV seropositive subjects enrolled for at least 6 months in an opiate agonist treatment (OAT) program will be referred to an off-site liver specialist.
  Then, 27 months of telemedicine: patients will be linked with the provider via two-way videoconferencing facilitated by an onsite case manager.
Period: Step 1: Months 0-9
Arm/Group | Sequence 1: 27 Month Usual Care, 9 Months Telemedicine | Sequence 2: 18 Month Usual Care, 18 Months Telemedicine | Sequence 3: 9 Months of Usual Care Followed by 27 Months Telemedicine
Started | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Completed | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Not Completed | 0; 0 Opioid Treatment Programs | 0; 0 Opioid Treatment Programs | 0; 0 Opioid Treatment Programs
Period: Step 2: Months 10-18
Arm/Group | Sequence 1: 27 Month Usual Care, 9 Months Telemedicine | Sequence 2: 18 Month Usual Care, 18 Months Telemedicine | Sequence 3: 9 Months of Usual Care Followed by 27 Months Telemedicine
Started | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Completed | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Not Completed | 0; 0 Opioid Treatment Programs | 0; 0 Opioid Treatment Programs | 0; 0 Opioid Treatment Programs
Period: Step 3: Months 19-27
Arm/Group | Sequence 1: 27 Month Usual Care, 9 Months Telemedicine | Sequence 2: 18 Month Usual Care, 18 Months Telemedicine | Sequence 3: 9 Months of Usual Care Followed by 27 Months Telemedicine
Started | 52; 4 Opioid Treatment Programs | 48; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Completed | 52; 4 Opioid Treatment Programs | 48; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Not Completed | 0; 0 Opioid Treatment Programs | 0; 0 Opioid Treatment Programs | 0; 0 Opioid Treatment Programs
Period: Period 4: Mos 28-36
Arm/Group | Sequence 1: 27 Month Usual Care, 9 Months Telemedicine | Sequence 2: 18 Month Usual Care, 18 Months Telemedicine | Sequence 3: 9 Months of Usual Care Followed by 27 Months Telemedicine
Started | 51; 4 Opioid Treatment Programs | 35; 4 Opioid Treatment Programs | 52; 4 Opioid Treatment Programs
Completed | 51; 4 Opioid Treatment Programs | 25; 4 Opioid Treatment Programs | 51; 4 Opioid Treatment Programs
Not Completed | 0; 0 Opioid Treatment Programs | 10; 0 Opioid Treatment Programs | 1; 0 Opioid Treatment Programs

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 312 | 290 | 602
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.94 (12.8) | 47.12 (13.1) | 48.06 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 115 | 233
  Male | 194 | 175 | 369
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 96 | 89 | 185
  Not Hispanic or Latino | 216 | 201 | 417
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 151 | 155 | 306
  Black/AA & Other | 161 | 135 | 296
Region of Enrollment [Number; unit: participants]
  United States | 312 | 290 | 602

OUTCOME MEASURES:

1. Primary Outcome: Observed Percentage of Patients in Both Arms Who Achieve Viral Eradication
Description: Percentage of patients who achieve viral eradication (defined as undetectable HCV RNA for 12 weeks post treatment cessation)
Time Frame: 12 weeks post treatment cessation
Population: Participants enrolled from 12 opioid treatment programs throughout New York State
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 312 | 290
Participants | 106 | 246

2. Secondary Outcome: Comparison of Treatment Initiation Percentages
Description: Comparison of treatment initiation percentages between the two arms, as measured by the percentage of patients that take an initial medication dose.
Time Frame: Up to 160 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 312 | 290
Participants | 126 | 268

3. Secondary Outcome: Comparison of Treatment Completion Rates
Description: Comparison of treatment completion percentages between the two arms.
Time Frame: Up to 210 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 312 | 290
Participants | 116 | 261

4. Secondary Outcome: Comparison of Patient Satisfaction
Description: We assessed patient satisfaction with healthcare delivery between the two arms through the Patient Satisfaction Questionnaire (PSQ) (1). The instrument is comprised of 18 questions from 7 subscales with responses on a 5-point Likert scale ranging from "1=Strongly Agree" to "5=Strongly Disagree". We administered the PSQ-18 at baseline and at the SVR time point. The higher the scored value, the higher the satisfaction. We calculated the score per participant, per time point, as the average of the scored values of all questions answered out of 18, and subsequently rounded the average score to the nearest integer (2).
  1. Marshall GN, Hays RD. The patient satisfaction questionnaire short-form (PSQ-18). Santa Monica, CA: RAND, 1994.
  2. Talal AH, Sofikitou EM, Wang K, Dickerson SS, Jaanimagi U, Markatou M. High Satisfaction with Patient-Centered Telemedicine for Hepatitis C Virus Delivered to Substance Users: A Mixed-Methods Study. Telemed J E-Health, 2023; 29: 395-407.
Time Frame: Baseline (initial time point) and at time HCV is cured, i.e., sustained virological response (up to 210 weeks).
Measure: Number; unit: % participants satisfied or high satisfy
Arm/Group | Control | Intervention
Number analyzed (Participants) | 106 | 238
% participants satisfied or high satisfy
  Initial Time point | 91.5 | 98.3
  HCV cure time point | 91.5 | 98.7

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire study period from screening through the two year post-treatment follow up perod.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 3/312 | 9/290
Serious Adverse Events (participants affected / at risk) | 0/312 | 0/290
Other Adverse Events (participants affected / at risk) | 0/312 | 0/290

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02933970/Prot_SAP_000.pdf